CLINICAL TRIAL: NCT01132248
Title: Activity of Mefloquine Against Urinary Schistosomiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Michael Ramharter, Ass. Prof. PD, Albert Schweitzer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDC-2010-1
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Schistosomiasis
Keywords: schistosomiasis, schistosoma haematobium
MeSH Terms: conditions — Schistosomiasis haematobia | interventions — Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mefloquine (Experimental): 15mg/kg mefloquine per dose Women receive two doses: One after the first trimester of pregnancy and the second at least one month after the first dose
  Interventions: Drug: Mefloquine
- S/P (Placebo Comparator): sulfadoxine-pyrimethamine IPTp will be administered following current WHO recommendations
  Interventions: Drug: S/P

INTERVENTIONS:
Drug: Mefloquine — 15mg/kg mefloquine per dose Women receive two doses: One after the first trimester of pregnancy and the second at least one month after the first dose
  Arms: Mefloquine
Drug: S/P — sulfadoxine-pyrimethamine IPTp will be administered following current WHO recommendations
  Arms: S/P

SUMMARY:
Urinary schistosomiasis is a debilitating disease in Central Africa and pregnant women are frequently suffering from this condition. Mefloquine is currently investigated as preventive treatment against malaria in pregnancy and mefloquine is also known to exert activity against schistosomiasis. The investigators want to test the hypothesis whether mefloquine may active against urinary schistosomiasis when used as preventive treatment against malaria in pregnancy.

DETAILED DESCRIPTION:
Objectives

The principal aim of this clinical trial is to evaluate whether mefloquine - when given as intermittent preventive treatment against malaria in pregnancy - shows in vivo activity against concomitant Schistosoma haematobium infection. This study is therefore a "proof of principle" study and is not intended to establish a clinically satisfying cure rate or to formally compare the efficacy of mefloquine with the standard therapy.

Hypothesis

Two underlying hypotheses have been formulated for this proof of principle study.

Primary hypothesis: Mefloquine reduces egg excretion of Schistosoma haematobium by 50% compared to sulfadoxine/pyrimethamine (S/P) treatment when given as IPTp Secondary hypothesis: Mefloquine may lead to an adequate cure rates of Schistosoma haematobium infections compared to S/P (>80%)

Trial Design

The evaluation of mefloquine activity against S. haematobium will be evaluated in the course of an open label multicenter randomized controlled trial assessing the efficacy, tolerability, and safety of mefloquine IPTp against malaria. This study is therefore a nested randomized controlled trial taking advantage of the randomization and treatment allocation procedures of the IPTp trial and assessing the additional efficacy outcome of reduction of S. haematobium egg excretion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women after first trimester and before 28th week of pregnancy
* HIV negative
* Egg excretion of Schistosoma haematobium (mean >10 eggs per mL urine)
* Asymptomatic (no signs of complicated Schistosomiasis, no severe anemia)
* Ability to comply with study protocol

Exclusion Criteria:

* Intake of anthelminthic or antimalarial drug within 2 months prior to inclusion
* Allergy to study drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reduction of egg excretion | 6 weeks after second IPTp
  Mefloquine reduces egg excretion of Schistosoma haematobium by 50% compared to sulfadoxine/pyrimethamine (S/P) treatment when given as IPTp

SECONDARY OUTCOMES:
Cure rate | 6 weeks after first and second IPTp
  Mefloquine may lead to an adequate cure rates of Schistosoma haematobium infections compared to S/P (>80%)

CONTACTS AND LOCATIONS:
Locations (2):
- Gabon (2):
  - Albert Schweitzer Hospital, Lambaréné, Moyen-Ogooué Province
  - Albert Schweitzer Hospital, Lambaréné

REFERENCES:
- [Derived] Salam RA, Das JK, Bhutta ZA. Effect of mass deworming with antihelminthics for soil-transmitted helminths during pregnancy. Cochrane Database Syst Rev. 2021 May 17;5(5):CD005547. doi: 10.1002/14651858.CD005547.pub4. PMID 33998661
- [Derived] Basra A, Mombo-Ngoma G, Melser MC, Diop DA, Wurbel H, Mackanga JR, Furstenau M, Zoleko RM, Adegnika AA, Gonzalez R, Menendez C, Kremsner PG, Ramharter M. Efficacy of mefloquine intermittent preventive treatment in pregnancy against Schistosoma haematobium infection in Gabon: a nested randomized controlled assessor-blinded clinical trial. Clin Infect Dis. 2013 Mar;56(6):e68-75. doi: 10.1093/cid/cis976. Epub 2012 Nov 21. PMID 23175561